CLINICAL TRIAL: NCT05201066
Title: An Open-label, Multicenter, Roll-over Study for Patients Who Have Completed a Prior Novartis-sponsored Sabatolimab (MBG453) Study and Are Judged by the Investigator to Benefit From Continued Treatment With Sabatolimab.
Brief Title: Roll-over Study for Patients Who Have Completed a Prior Novartis-sponsored Sabatolimab (MBG453) Study and Are Judged by the Investigator to Benefit From Continued Treatment With Sabatolimab.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453B12206B; 2021-004422-30 (EudraCT Number); 2024-515281-14-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2022-01-03; First posted 2022-01-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic
Keywords: roll-over study; MBG453; sabatolimab; azacitidine; decitabine; venetoclax; spartalizumab; HMA; INQOVI (oral decitabine)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Decitabine; spartalizumab; sabatolimab; Azacitidine; venetoclax; decitabine and cedazuridine drug combination

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- sabatolimab + azacitidine (Experimental): Patients will take sabatolimab 800 mg i.v and azacitidine 75 mg/m2/d d1-7 s.c. or i.v./q4w or sabatolimab 400 mg i.v/q2w and azacitidine 75 mg/m2/d d1-7 s.c. or i.v./q4w.
  Interventions: Drug: sabatolimab; Drug: azacitidine
- sabatolimab + decitabine (Experimental): Patients will take Sabatolimab 400 mg i.v/q2w and decitabine 20 mg/m2/d d1-5 i.v.
  Interventions: Drug: decitabine; Drug: sabatolimab
- sabatolimab + venetoclax + azacitidine (Experimental): Patients will take sabatolimab 200 mg i.v./q2w and venetoclax 400 mg p.o. d1-14/q4wk and azacitidine 75 mg/m2/d d1-7/q4w.
  Interventions: Drug: sabatolimab; Drug: azacitidine; Drug: venetoclax
- sabatolimab + spartalizumab + decitabine (Experimental): Patients will take sabatolimab 400 mg i.v./q2w and decitabine 20 mg/m2/d d1-5 i.v. and spartalizumab 100 mg i.v/q2w.
  Interventions: Drug: decitabine; Drug: spartalizumab; Drug: sabatolimab
- sabatolimab + HMA (Experimental): Patients will take sabatolimab 800 mg and azacitidine 75 mg/m2/d d1-7 or decitabine 20 mg/m2/d d1-5/ all q4w
  HMA means hypomethylating agents. Hypomethylating agents are azacitidine and decitabine.
  Interventions: Drug: sabatolimab; Drug: INQOVI (oral decitabine)
- sabatolimab (Experimental): Patients will take sabatolimab 800 mg i.v q4w.
  Interventions: Drug: sabatolimab

INTERVENTIONS:
Drug: decitabine — Solution for intravenous infusion
  Arms: sabatolimab + decitabine; sabatolimab + spartalizumab + decitabine
Drug: spartalizumab — Solution for intravenous infusion
  Other Names: PDR001
  Arms: sabatolimab + spartalizumab + decitabine
Drug: sabatolimab — Solution for intravenous infusion
  Other Names: MBG453
Drug: azacitidine — Solution for subcutaneous injection or intravenous infusion
  Arms: sabatolimab + azacitidine; sabatolimab + venetoclax + azacitidine
Drug: venetoclax — Tablet for oral administration
  Arms: sabatolimab + venetoclax + azacitidine
Drug: INQOVI (oral decitabine) — Tablet for oral administration. HMA = azactidine or decitabine INQOVI = decitabine (oral)
  Arms: sabatolimab + HMA

SUMMARY:
This study is intended to collect safety data from participants who completed the parent protocols but are still benefiting from study treatment. The study population consists of participants who tolerate study treatment of the parent studies. Collecting safety information from long-term exposure might offer the unique opportunity to detect rare Adverse Events.

DETAILED DESCRIPTION:
This is a multicenter, open label, roll-over study to collect and assess safety of sabatolimab in participants who are treated in current Novartis-sponsored parent studies and who are benefiting from continued study treatment including sabatolimab as judged by the investigator.

There is no conventional screening period in this study as participants are expected to transition directly from treatment on the parent protocol to treatment on this roll-over protocol. Participants who are candidates for the roll-over protocol will be evaluated by the investigator in the parent protocol for eligibility for the roll-over protocol. If eligible, the parent protocol end of treatment visit will be performed and the informed consent for the roll-over protocol will be signed. Participants then continue treatment on this protocol with the next planned dose of sabatolimab as monotherapy or with other combination agent(s).

The treatment with sabatolimab and combination agent(s), as applicable, is continued according to the schedule in the parent study. Adverse events (AEs) will be collected continuously throughout the study and participants will be questioned about adverse events at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is currently enrolled in a Novartis-sponsored study with sabatolimab, is being treated with sabatolimab, and has fulfilled all requirements in the parent study.
2. Participant is currently benefiting from the treatment with sabatolimab as determined by guidelines of the parent protocol and investigator's judgment.
3. Participant has demonstrated compliance, as assessed by the investigator, with the parent study protocol requirements.
4. Willingness and ability to comply with scheduled visits, treatment plan and any other study procedures.
5. Written informed consent obtained prior to enrolling in the roll-over study.

Exclusion Criteria:

1. Participants in cohorts or treatment groups not receiving sabatolimab in the parent protocol.
2. Participant has been permanently discontinued from sabatolimab treatment in the parent study due to unacceptable toxicity, non-compliance to study procedures, withdrawal of consent or any other reason.
3. Participant currently has unresolved toxicities for which sabatolimab dosing has been interrupted in the parent study (participants meeting all other eligibility criteria may be enrolled once toxicities have resolved to allow sabatolimab dosing to resume).
4. Pregnant or nursing (lactating) women. Where pregnancy is defined as the state of a female after conception confirmed by a positive serum hCG laboratory test and until the termination of gestation.
5. Participant not willing to comply with the contraception requirements outlined in the exclusion criteria of the parent protocol.
6. Local access to commercially available sabatolimab for parent protocol indications.

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2028-02-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | 5 years
  An AE is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study. An AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  An SAE is defined as any adverse event [appearance of (or worsening of any pre-existing)] undesirable sign(s), symptom(s), or medical conditions(s) which meets any one of the following criteria: fatal, life-threatening, results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, may have caused a congenital anomaly/birth defect, requires intervention to prevent permanent impairment or damage.
Severity of AEs and SAEs | 5 years
  Severity of AEs and SAEs will be measured according to the CTCAE v5.0

SECONDARY OUTCOMES:
Duration of exposure to sabatolimab | 5 years
  The length of time patients will be exposed to sabatolimab and will be reported by treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (2):
  - Oregon Health Sciences University, Portland, Oregon
  - Huntsman Cancer Institute Univ of Utah, Salt Lake City, Utah
- Novartis Investigative Site, Clayton, Victoria, Australia
- Novartis Investigative Site, Florianópolis, Santa Catarina, Brazil
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- China (2):
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Tianjin
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Toulouse, France
- Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Greece (2):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Pátrai
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Novartis Investigative Site, Fukushima, Japan
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Spain (3):
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com